CLINICAL TRIAL: NCT01630538
Title: Phase II Pilot Study of Cyclophosphamide Therapy for Refractory Antibody-Mediated Rejection in Kidney Transplantation
Brief Title: Cyclophosphamide Therapy for Refractory Antibody-Mediated Rejection (AMR) in Kidney Transplants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After March 2015, unable to enroll due to patients meeting exclusion criteria.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMCT-01
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Antibody Mediated Rejection
Keywords: Transplantation
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide (Experimental): Cyclophosphamide 1.5 mg/kg orally daily for 180 days (26 weeks) adjusted for renal function.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 1.5 mg/kg orally daily for 180 days adjusted for renal function
  Other Names: Procytox

SUMMARY:
The study hypothesis is that short-term low dose cyclophosphamide therapy will be effective in resolving inflammation in patients with late phase antibody-mediated rejection refractory to current standard of care treatment.

DETAILED DESCRIPTION:
There is no consensus on the optimal treatment of de novo donor specific antibody-mediated rejection. Optimizing baseline immunosuppression (calcineurin inhibitor (CNI), anti-proliferative agent, and anti-inflammatory) is considered foundational but is insufficient. Pulse steroids are routinely used. A number of immunosuppressive approaches have been tried in uncontrolled trials. The strongest evidence, at least for early antibody-mediated rejection (< 6 months from transplant), exists for plasmapheresis, with or without low dose IVIg, or high dose IVIg alone. However, as noted in a recent FDA workshop, "while the literature suggests that [these agents] have evidence of efficacy for the management of acute antibody-mediated rejection, and could be considered as standard of care, treatment regimes have not been standardized or optimized." Moreover the evidence supporting efficacy of this approach in late, as opposed to early antibody-mediated rejection is distinctly lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a living or deceased donor kidney transplant
* Failed current standard of care for late antibody-mediated rejection
* Persistent de novo donor specific antibody and a concurrent biopsy with histologic evidence of acute antibody-mediated inflammation
* Adults with reproductive potential must agree to use approved methods of birth control while in the study

Exclusion Criteria:

* Leukopenia (WBC) < 3.0 x 109/L
* Creatinine Clearance less than or equal to 25 ml/min/1.73m2
* HCV or HBV positive
* BKV or CMV viremia assessed by PCR
* Any active infection
* Use of other investigational drugs within 4 weeks of study
* Pregnancy/breast feeding/unwilling or unable to take birth control
* Active malignancy
* de novo DSA occurring equal to or greater than15 years after kidney transplant
* Screening biopsy with equal to or greater than cg2 on Banff criteria
* Cumulative/lifetime dose of cyclophosphamide, including anticipated total study dose (calculated according to Creatinine Clearance and mg/kg/day) equal to or greater than 36 g.
* Any condition that, in the opinion of the investigator, would pose risk to the subject's safe participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Microvascular inflammation | month 6
  Histologic resolution of acute antibody-mediated inflammation in a 6 month post-treatment biopsy (Banff histology scores: g, v, ptc, C4d +ve)

SECONDARY OUTCOMES:
titre of donor specific antibody (DSA) | 6 and 12 months
  Change in the level of de novo DSA between enrolment and at 6 and 12 months post-enrollment
antibody-mediated tissue injury | month 6
  Change in antibody-mediated tissue injury between the enrollment and post-treatment kidney transplant biopsy samples
Urine Albumin/Creatinine ratios | month 6 and 12
  Change in urine albumin/creatinine ratio between enrolment and 6 and 12 month post-enrolment samples
Creatinine Clearance and estimated GFR | month 6 and 12
  Evaluation of Creatinine Clearance, and estimated GFR using the Chronic Kidney Disease Epidemiology (CKR-EPI) equation
Graft Survival | month 6 and 12
Patient Survival | month 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Nickerson, MD, Principal Investigator — University of Manitoba; David N Rush, MD, Study Chair — University of Manitoba
Locations (1):
- Transplant Manitoba Adult Kidney Transplant Program, Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Karpinski M, Ho J, Storsley LJ, Goldberg A, Birk PE, Rush DN, Nickerson PW. Evolution and clinical pathologic correlations of de novo donor-specific HLA antibody post kidney transplant. Am J Transplant. 2012 May;12(5):1157-67. doi: 10.1111/j.1600-6143.2012.04013.x. Epub 2012 Mar 19. PMID 22429309
- [Background] Archdeacon P, Chan M, Neuland C, Velidedeoglu E, Meyer J, Tracy L, Cavaille-Coll M, Bala S, Hernandez A, Albrecht R. Summary of FDA antibody-mediated rejection workshop. Am J Transplant. 2011 May;11(5):896-906. doi: 10.1111/j.1600-6143.2011.03525.x. PMID 21521465